CLINICAL TRIAL: NCT06778226
Title: ThRombectomy In Mild Ischemic Stroke With a Visible Intracranial veSsel Occlusion
Acronym: TRIMIS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Brown University (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Negar Asdaghi, Associate Professor of Neurology, University of Miami
Other Study IDs: 20180038
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Immediate Endovascular Therapy: Data previously collected from medical records will be analyzed with the purpose of studying the efficiency of Immediate Endovascular Therapy. Length of the cohort is 6 years.
- Delayed Endovascular Therapy: Data previously collected from medical records of participants will be analyzed with the purpose of studying the efficiency of Delayed Endovascular Therapy. Length of the cohort is 6 years.
- Medical Management: Data previously collected from medical records of participants will be analyzed with the purpose of studying the efficiency of Medical Management. Length of the cohort is 6 years.

SUMMARY:
The purpose of TRIMIS is to study how a medical procedure by the name of endovascular therapy compares to medical treatment alone in patients with mild stroke and a blood vessel occlusion in the brain

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke in an adult patient (18 years of age or older).
2. Onset (Last Seen Normal) time to treatment time <24 hours or unknown Last Seen Normal in whom Endovascular Therapy could be considered per local radiographic guidelines.
3. Mild stroke defined as an NIH Stroke Scale ≤ 5 at the time of treatment decision.

   a. Patients with NIH Stroke Scale=0 can be included in the study if they have relevant abnormalities on neurological exam.
4. An acute intracranial vessel occlusion (Intracranial Internal Carotid Artery terminus (T or L clot), Middle Cerebral Artery (M1, M2, M3/beyond), Anterior Cerebral Artery (A1, A2, A3), V4, Basilar, Posterior Cerebral Artery) defined by non-invasive acute imaging (Computed Tomography, angiography (Computed Tomography Angiography) or Magnetic Resonance angiography (MRA)) that is neurologically relevant to the presenting symptoms and signs.

Exclusion Criteria:

1. Stroke symptoms due to another non-ischemic acute neurological condition such as seizure with Post-ictal Todd's paralysis or focal neurological signs due to severe hypo- or hyperglycemia.
2. Hyperdensity on Non-contrast Computed Tomography consistent with intracranial hemorrhage. Any clinical suspicion of any intracranial hemorrhage even in the absence of visible blood on baseline brain imaging.
3. Large acute stroke >1/3 Middle Cerebral Artery territory or Alberta Stroke Programme Early CT score (ASPECTS<6 or established frank hypodensity relevant to the presenting acute stroke already visible on baseline CT scan.
4. Findings on acute CT or MRI to suggest that the
5. Patient has a severe or fatal or disabling illness that will impact decision regarding acute reperfusion therapies.
6. Pregnancy.
7. Clinical history, past imaging and clinical judgment suggest that the intracranial occlusion is chronic.
8. Stroke occurred as an inpatient.
9. Inclusion into any randomized control trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute stroke patients treated at participating sites in North America, South America, Europe, Asia, and Australia.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90 Days
  Scores range from 0-6. (0 = normal, 6 = dead).

SECONDARY OUTCOMES:
Symptomatic Intracerebral Hemorrhage (sICH) | 48 hours
  Scores range from 0-3, higher scores indicate worse outcomes
Change in National Institute of Health Stroke Scale (NIHSS) | 24 hours, 7 days
  Scores range 0-42; higher scores indicate worse outcomes
Modified Rankin Scale | 7 days
  Scores range from 0-6. (0 = normal, 6 = dead).

CONTACTS AND LOCATIONS:
Overall Officials: Negar Asdaghi, MD, Principal Investigator — University of Miami; Shadi Yaghi, MD, Principal Investigator — Brown University; Thanh Nguyen, MD, Principal Investigator — Boston Medical Center
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No